CLINICAL TRIAL: NCT07398937
Title: A Randomized, Open-label, Multicenter Phase II Clinical Trial Evaluating the Efficacy and Safety of Serplulimab Combined With Chemotherapy Versus Nivolumab Combined With Chemotherapy as Neoadjuvant Therapy in Resectable Stage II-IIIa Squamous NSCLC.
Brief Title: Comparison of Serplulimab Versus Nivolumab in Neoadjuvant Therapy for Resectable Stage II-IIIA Squamous NSCLC
Acronym: ECTOP-1036
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT314
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Resectable Stage II-IIIa Squamous NSCLC
Keywords: lung cancer; immunotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Drug Therapy; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serplulimab + chemotherapy (Experimental): Serplulimab injection [300 mg, administered on Day 1, Q3W (once every 3 weeks)] + paclitaxel (albumin-bound) for injection [260 mg/m2, highest dose Not More Than 400 mg, administered on Day 1, Q3W] + carboplatin injection (AUC=5, highest dose Not More Than 750 mg, administered on Day 1, Q3W) for 2-3 cycles;
  Interventions: Drug: Serplulimab + chemotherapy
- Nivolumab + chemotherapy (Active Comparator): Nivolumab [360 mg, administered on Day 1, Q3W (once every 3 weeks)] + paclitaxel (albumin-bound) for injection [260 mg/m2, highest dose Not More Than 400 mg, administered on Day 1, Q3W] + carboplatin injection (AUC=5, highest dose Not More Than 750 mg, administered on Day 1, Q3W) for 2-3 cycles;
  Interventions: Drug: Nivolumab + chemotherapy

INTERVENTIONS:
Drug: Serplulimab + chemotherapy — Serplulimab injection [300 mg, administered on Day 1, Q3W (once every 3 weeks)] + paclitaxel (albumin-bound) for injection [260 mg/m2, highest dose Not More Than 400 mg, administered on Day 1, Q3W] + carboplatin injection (AUC=5, highest dose Not More Than 750 mg, administered on Day 1, Q3W) for 2-3 cycles
  Arms: Serplulimab + chemotherapy
Drug: Nivolumab + chemotherapy — Nivolumab [360 mg, administered on Day 1, Q3W (once every 3 weeks)] + paclitaxel (albumin-bound) for injection [260 mg/m2, highest dose Not More Than 400 mg, administered on Day 1, Q3W] + carboplatin injection (AUC=5, highest dose Not More Than 750 mg, administered on Day 1, Q3W) for 2-3 cycles;
  Arms: Nivolumab + chemotherapy

SUMMARY:
This trial is a randomized, controlled, multicenter, open-label study, planning to enroll 116 subjects with resectable stage II-IIIa squamous NSCLC confirmed by histopathology or cytology, aiming to evaluate the efficacy and safety of serplulimab compared to nivolumab combined with chemotherapy in neoadjuvant therapy. This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1036.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years at time of study entry.
2. The International Federation of Gynecology and Obstetrics (FIGO) 2018 Stages II-IIIA squamous non-small cell lung cancer confirmed by histopathology or cytology.
3. The patient with stage II-IIIA squamous non-small cell lung cancer confirmed by histopathology or cytology;
4. Able to tolerate complete lung cancer resection;
5. WHO/ECOG performance status of 0 or 1.

Exclusion Criteria:

1. Other pathological histological types of non-small cell lung cancer subjects, including adenocarcinoma subjects, squamous-adenocarcinoma mixed cancer subjects, and NSCLC containing components of small cell lung cancer and neuroendocrine carcinoma.
2. EGFR sensitivity mutation or ALK, ROS1 gene rearrangement;
3. Known severe allergy to any components of carboplatin/albumin paclitaxel and other drugs;
4. Central nervous system (CNS) or leptomeningeal metastases confirmed by imaging or pathology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission (PCR) rate | From randomization up to a median of 30 months after randomization
  Pathologic complete response (pCR) rate is defined as the number of randomized participants with absence of residual tumor in lung and lymph nodes as evaluated by investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No